CLINICAL TRIAL: NCT03295890
Title: Dry Needling on the Treatment of Chronic Somatosensory Tinnitus: An Open Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: USaoPauloGHGZ
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Tinnitus; Trigger Point Pain, Myofascial; Somatosensory Disorders
Keywords: myofascial trigger point, tinnitus, dry needling
MeSH Terms: conditions — Tinnitus; Myofascial Pain Syndromes; Somatosensory Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Needling (Sham Comparator): Intervention = Sham Needling
  Interventions: Procedure: Dry Needing
- Active Needling (Active Comparator): Intervention = Active Needling
  Interventions: Procedure: Dry Needing

INTERVENTIONS:
Procedure: Dry Needing — Dry Needling

SUMMARY:
Self paring study, double blind placebo controlled with chronic tinnitus patients attended at the Tinnitus Research Group HC- FMUSP, complaining of neck and/or cervical pain and with myofascial trigger point in the head, neck and/or shoulder. They were submitted to a complete otolaryngologist evaluation which included history, physical examination and myofascial trigger point checkup. Patients also performed blood tests, tonal and vocal audiometry, and psychoacoustic tinnitus measures. Self paring study, double blind placebo controlled. Each patient will be subjected to the dry needling placebo, 4 sessions, 1 per week, with placebo stretching, followed by washout period of two weeks, and 4 more dry needling therapeutic sessions and active stretching. On the first day of the study will be conducted the following evaluation: questionnaires THI and NDI, quantification of cervical pain and tinnitus through the Visual analogue scale (VAS), search and confirmation of the presence of PGM and cervical pain, psychoacoustic measures and somatic tests. This evaluation will be repeated at the end of the four placebo sessions, at the beginning of therapeutic needling sessions and at the end of the same.

DETAILED DESCRIPTION:
The first phase of the study will be the placebo needling, performed with a sham needle and following the same procedures than the therapeutic treatment. Four placebo sessions will be performed, 1 per week, with placebo stretching, followed by washout period of two weeks, and 4 more dry needling therapeutic sessions, also once a week and active stretching. The muscles selected for dry needling were frontal, temporal, trapezius, masseter, sternocleidomastoid (SCM), head splenius, scalene, medial pterygoid, lateral pterygoid, rhomboid.

Procedure technique Each patient was recommended to assume a relaxed posture suitable to access the muscles being treated, instructed to expose the painful area, settled himself in supine, prone, or side lying positions, at a stretcher or a chair, depending on the muscle to be treated. The main therapist performed MTP target with a pen, hands antisepsis, gloves wear and skin area cleaning with 70% isopropyl alcohol prior to needling. Along all procedure the main therapist was able to view the patient's face and to receive regular treating feedback. A sterile disposable filament needle was inserted directly perpendicular through the skin using a guide tube that was then removed. Depth needle penetration with slow sidelong direction in and outside displacements were performed through the muscle until reach MTP spot. The patient's reaction indicated a "DEQI" (name given for the vague sensation of needle-specific pain) or a "twitch response" (deflagration of a contractile muscle answer in the moment that maximum muscle shortening fibers were broken). At this point needle was leaved static in situ for 30-60 seconds. After the correct treatment needle was removed and the muscle was active stretched.

Variables studied before and after therapeutic needling were:

1. Tinnitus annoying as measured by AVS.
2. Pain magnitude as measured by AVS.
3. Tinnitus impact on patient's quality of life through THI questionnaire validated for Portuguese language.
4. Cervical pain impact on patient's quality of life through NDI questionnaire validated for Portuguese language.
5. Tinnitus MML through psychoacoustic measures.

ELIGIBILITY:
Inclusion Criteria:

* With constant tinnitus, unilateral or bilateral, for more than 6 months,
* Both sexes,
* Over 18 years,
* Presence of at least one PGM (active or latent),
* Diagnosis of Myofascial pain syndrome, according to the criteria of Travell and Simons.

Exclusion Criteria:

* With prior experience with the use of needles for therapeutic purposes,
* With formal contraindication to dry needling, as chronic use of anticoagulants or hematologic diseases,
* Those who refuse the proposed therapies, for example, phobia of needles,
* In use of medications for pain able to interfere with the result of the study, such as anti-inflammatory and or muscle relaxers, until 30 days before the initial assessment,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07-29 (Actual); Primary Completion 2018-06-05 (Estimated); Study Completion 2020-07-29 (Estimated)

PRIMARY OUTCOMES:
Placebo Dry Needling | 4 weeks
  Placebo Needling on trigger points

SECONDARY OUTCOMES:
Active Dry needling | 4 weeks
  Therapeutic needling on trigger points

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Bento, MD PhD, Study Chair — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No